CLINICAL TRIAL: NCT04079608
Title: Rigorous Evaluation of High School FLASH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ETR Associates (Other)
Collaborators: Public Health Seattle King County (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FLASH study
Record Dates: First submitted 2019-09-03; First posted 2019-09-06 (Actual); Last update posted 2019-09-11 (Actual); Status verified 2019-09

CONDITIONS: Pregnancy Related; Sexual Behavior; STD
Keywords: Pregnancy; Adolescents; STD; Decision making; Harm reduction; Prevention education
MeSH Terms: conditions — Sexual Behavior; Harm Reduction | interventions — Sex Education

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FLASH curriculum (Experimental): Students who will receive the FLASH high school curriculum.
  Interventions: Behavioral: FLASH curriculum
- Sexual Health Education for Adolescents (Active Comparator): Students will receive a five-session knowledge-based sexual health curriculum designed for classroom settings.
  Interventions: Behavioral: Sexual Health Education for Adolescents

INTERVENTIONS:
Behavioral: FLASH curriculum — High School FLASH is a 15-session comprehensive sexual health curriculum designed for classroom settings in grades 9 to 12. The basis of High School FLASH is a public health approach to behavior change. The primary strategy used in the FLASH curriculum for preventing teen pregnancy, sexually transmitted diseases (STDs), and sexual violence is to address student behaviors and attitudes. To this end, FLASH uses a harm reduction and behavior change framework, implements best practices as outlined in the research on effective programs, addresses risk and protective factors for program goals, and rests on the theory of planned behavior. The instructional approach of High School FLASH employs key concepts in every lesson, which enables teachers to hone in on the risk and protective factors outlined in the curriculum logic model.
  Arms: FLASH curriculum
Behavioral: Sexual Health Education for Adolescents — Sexual Health Education for Adolescents is a five-session knowledge-based sexual health curriculum designed for classroom settings. The lessons cover the reproductive system, pregnancy, birth control, abstinence, human immunodeficiency virus (HIV) and other sexually transmitted diseases (STDs), and healthy relationships. The goal of the curriculum is to increase student knowledge in all content areas. The primary strategy employed by Sexual Health Education for Adolescents is to address the cognitive learning domain. The curriculum aligns to national health education standards and is intended to be implemented by classroom teachers. The lessons can be delivered according to the schedule that works best for schools (e.g., twice a week, once a week, every days) within a school semester.
  Arms: Sexual Health Education for Adolescents

SUMMARY:
High School FLASH is a 15-session comprehensive sexual health curriculum designed for classroom settings in grades 9 to 12. The basis of High School FLASH is a public health approach to behavior change. The primary strategy used in the FLASH curriculum for preventing teen pregnancy, sexually transmitted diseases (STDs), and sexual violence is to address student behaviors and attitudes. To this end, FLASH uses a harm reduction and behavior change framework, implements best practices as outlined in the research on effective programs, addresses risk and protective factors for program goals, and rests on the theory of planned behavior. The instructional approach of High School FLASH employs key concepts in every lesson, which enables teachers to hone in on the risk and protective factors outlined in the curriculum logic model. The curriculum covers the following topics: reproductive system, pregnancy, sexual orientation and gender identity, healthy relationships, coercion and consent, online safety, abstinence, birth control, preventing human immunodeficiency virus (HIV) and other STDs, condoms, STD testing, communicating and decision making, and improving school health. The curriculum aligns with national health education standards.

DETAILED DESCRIPTION:
High School FLASH is a 15-session comprehensive sexual health curriculum designed for classroom settings in grades 9 to 12. The basis of High School FLASH is a public health approach to behavior change. The primary strategy used in the FLASH curriculum for preventing teen pregnancy, sexually transmitted diseases (STDs), and sexual violence is to address student behaviors and attitudes. To this end, FLASH uses a harm reduction and behavior change framework, implements best practices as outlined in the research on effective programs, addresses risk and protective factors for program goals, and rests on the theory of planned behavior. The instructional approach of High School FLASH employs key concepts in every lesson, which enables teachers to hone in on the risk and protective factors outlined in the curriculum logic model. The curriculum covers the following topics: reproductive system, pregnancy, sexual orientation and gender identity, healthy relationships, coercion and consent, online safety, abstinence, birth control, preventing human immunodeficiency virus (HIV) and other STDs, condoms, STD testing, communicating and decision making, and improving school health. The curriculum aligns with national health education standards. FLASH is ideally taught 2-5 times per week for 15 sessions lasting 50 minutes, or 10 sessions lasting 70-80 minutes, covering the same content. The curriculum is designed to be flexible to ensure sustainability in a variety of school environments.

The counterfactual condition is called Sexual Health Education for Adolescents, which is a five-session knowledge-based sexual health curriculum designed for classroom settings. The lessons cover the reproductive system, pregnancy, birth control, abstinence, HIV and other STDs, and healthy relationships. The goal of the curriculum is to increase student knowledge in all content areas. The primary strategy employed by Sexual Health Education for Adolescents is to address the cognitive learning domain. The curriculum aligns to national health education standards and is intended to be implemented by classroom teachers. The lessons can be delivered according to the schedule that works best for schools (e.g., twice a week, once a week, every days) within a school semester.

Students were recruited from 9th (South) or 10th (Midwest) grade health classes. The research team met with district and school administrators and health teachers to explain the study, data collection processes, and to answer questions. The FLASH study enrolled students from required health classes from 20 schools in the South and the Midwest. In the Midwest, we worked with two districts; one of the districts contributed 9 of the 10 high schools and the other district contributed one high school to the evaluation study. In the South, we have partnered with 10 schools in 5 counties, representing 5 different districts. One of these districts contributed 6 schools to the evaluation study and the remaining 4 districts each contributed 1 high school to the study.

Randomization was staggered and rolled-out by region to ensure that implementation started at the same time for all schools but only started in one region at a time. School enrollment was used as a stratification variable, so that schools assignments to the intervention and control arm were balanced within stratum. Randomization was performed within each region at the school level and was stratified into two categories by school size. For the Midwest region, small was defined as <500 enrollment and large was =>1000. For the Southern region, small was defined as <700 enrollment and large was =>700.

Active parental consent and student assent were obtained prior to any data collection. The steps in the consent process are discussed below:

1. Two weeks or more prior to the surveys (as determined by the participating schools), evaluation staff went to each participating health class and provided an overview of the study and distributed parent consent forms to all students in the class, requesting that they take them home to their parents for review and return the signed forms to their classroom teacher with parents' decisions regarding participation marked on the form. In the Southern schools, students received a gift card worth $10 for returning parent consent forms. The Midwestern schools' administration would not allow for the distribution of any type of incentives; thus, these schools received a class reward for taking part in the parent consent process and reaching a threshold (e.g., 75% or more of students return parent consent regardless of whether parents say "yes" or "no"). All consent forms were translated into languages requested by each district.
2. Evaluation staff returned multiple times (e.g., 2-3) during the collection period as agreed upon with the classroom teacher to check on the parent consent return rates and did brief reminders to students.
3. Between evaluation staff visits to the classrooms, teachers were asked to remind students to return parent consent forms daily over the collection period and provided additional forms to students who needed them.
4. After two weeks, evaluation staff worked with the schools to make calls to parents using a scripted protocol to read the consent form over the phone and secure parents' decisions or send them the form for them to return it by mail with their decision. In nine schools within one district in the Midwest region, we trained their nursing office staff (which included Health Educational Assistants and Licensed Practical Nurses) to make verbal consent calls home to parents at the request of district administration. These staff members are already responsible for communicating with parents about health-related matters and given that this was a health-related research study, the administration felt that these calls would be better received by their staff, rather than unfamiliar data collectors.

The primary source of data for the outcome analyses is the student self-report survey. The survey was administered three times over the course of the study. In the Midwest region this occurred: Fall 2016 (baseline), Spring 2017 (3-month follow-up), and Fall-Winter 2017-2018 (12-month follow-up). In the Southern region, data collection took place: Fall 2017 (baseline), Spring 2018 (3-month follow-up) and Fall-Winter 2018-2019 (12-month follow-up). Data were collected by trained data collectors in schools using handheld tablets. For students who left school after baseline but before follow-up surveys could be administered, we worked to survey these students at their new schools, online, or by mail.

ELIGIBILITY:
Inclusion criteria was determined at three levels:

* District level eligibility: Districts must have been from regions with teen birth rates at or above the national average at the time of study recruitment. They also much have agreed with randomization of mainstream schools to either High School FLASH or the five-session knowledge-based comparison condition. We worked with 7 different districts in two different regions of the U.S. - the Midwest (2 districts) and the South (5 districts).
* School level eligibility: Schools were eligible to participate if they: (1) agreed with inviting all students in targeted grade level in the fall semester required class to take part in the study (9th or 10th grades depending on health education course placement); (2) had a policy environment that enabled implementation of all FLASH components if randomized to intervention condition; (3) were in a district not currently mandating comprehensive sexuality education or using an evidence-based sexual health curriculum in school or for after-school programs; and (4) have schools large enough to ideally contribute 40 or more students to the study.
* Student level eligibility: Student enrollment into the study must have included (1) being in targeted classes during the enrollment window (fall semester 2016 in the Midwest and fall semester 2017 in the South), (2) providing positive parent consent to take part in study survey; and (3) providing assent to take part in the survey.

Exclusion Criteria:

* Anyone not meeting inclusion criteria

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1597 (Actual)
Dates: Start 2016-10-05 (Actual); Primary Completion 2019-01-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Self-reported rates of vaginal sex | 3 months post-intervention
  Measured with a single item required and provided by the funder: "In the past 3 months, have you had vaginal intercourse, even once?" Yes/No
Self-reported rates of vaginal sex | 12 months post-intervention
  Measured with a single item required and provided by the funder: "In the past 3 months, have you had vaginal intercourse, even once?" Yes/No
Self-reported rates of vaginal sex without a condom or other birth control | 3 months post-intervention
  Combined the following two questions required and provided by the funder: "In the past 3 months, have you had vaginal intercourse without you or your partner using a condom?" and "In the past 3 months, how many times have you had vaginal intercourse without you or your partner using any of these methods of birth control: birth control pills, the shot, the patch, the ring, intrauterine device (IUD), or Implant" New outcome was coded 'yes' if either question was endorsed and 'no' if both questions were responded to as 'no'
Self-reported rates of vaginal sex without a condom or other birth control | 12 months post-intervention
  Combined the following two questions required and provided by the funder: "In the past 3 months, have you had vaginal intercourse without you or your partner using a condom?" and "In the past 3 months, how many times have you had vaginal intercourse without you or your partner using any of these methods of birth control: birth control pills, the shot, the patch, the ring, intrauterine device (IUD), or Implant" New outcome was coded 'yes' if either question was endorsed and 'no' if both questions were responded to as 'no'

SECONDARY OUTCOMES:
Self-reported initiation of vaginal sex | 3 months post-intervention
  Measured with a single item required and provided by the funder: "Have you ever had vaginal sex?" Coding is 0 = 'no', 1 = 'yes'. This will only be analyzed on subjects reporting no to this same question at baseline.
Self-reported initiation of vaginal sex | 12 months post-intervention
  Measured with a single item required and provided by the funder: "Have you ever had vaginal sex?" Coding is 0 = 'no', 1 = 'yes'. This will only be analyzed on subjects reporting no to this same question at baseline.
Self-reported knowledge of sexually transmitted disease (STD) testing | 3 months post-intervention
  There are three knowledge measures developed specifically for this study around STD testing. "Have you heard of a clinic or doctor in your community where teens can get sexual health information and tests?" Coded 'yes', 'no', and 'not sure'. "If you needed to be tested, how comfortable would you be going to a clinic to be tested for STDs and HIV?" and "Imagine you or a friend wanted to get an STD test. How sure are you that you could go or help a friend to go to a clinic and get it?" both coded using a 4 point scale ranging from 'Very sure' or 'Very comfortable' to 'Not sure at all' or 'Not at all comfortable'.
Self-reported knowledge of sexually transmitted disease (STD) testing | 12 months post-intervention
  There are three knowledge measures developed specifically for this study around STD testing. "Have you heard of a clinic or doctor in your community where teens can get sexual health information and tests?" Coded 'yes', 'no', and 'not sure'. "If you needed to be tested, how comfortable would you be going to a clinic to be tested for STDs and HIV?" and "Imagine you or a friend wanted to get an STD test. How sure are you that you could go or help a friend to go to a clinic and get it?" both coded using a 4 point scale ranging from 'Very sure' or 'Very comfortable' to 'Not sure at all' or 'Not at all comfortable'.
Self-reported comfort with family communication regarding sexual health | 3 months post-intervention
  This is measured using the following two questions developed specifically for this study: "How comfortable are you talking about relationships, sexual health, or sex with your mother or female guardian?" "How comfortable are you talking about relationships, sexual health, or sex with your father or male guardian?" Coded 1 = 'comfortable', 2 = 'not comfortable'
Self-reported comfort with family communication regarding sexual health | 12 months post-intervention
  This is measured using the following two questions developed specifically for this study: "How comfortable are you talking about relationships, sexual health, or sex with your mother or female guardian?" "How comfortable are you talking about relationships, sexual health, or sex with your father or male guardian?" Coded 1 = 'comfortable', 2 = 'not comfortable'

CONTACTS AND LOCATIONS:
Overall Officials: Karin Coyle, PhD, Principal Investigator — ETR
Locations (1):
- ETR, Scotts Valley, California, United States